CLINICAL TRIAL: NCT04836507
Title: An Open-label, Multi-center, Single-arm Phase 1/2 Study to Assess Tolerability, Safety and Efficacy of CRC01 in Adult Patients With Relapsed or Refractory Large B-cell Lymphoma
Brief Title: Study of Efficacy and Safety of CRC01 in Adult Large B-cell Lymphoma Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Curocell Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC01-01
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Relapsed Large B-cell Lymphoma; Refractory Large B-cell Lymphoma; Diffuse Large B-cell Lymphoma (DLBCL); Primary Mediastinal Large B-Cell Lymphoma (PMBCL); High-grade B-cell Lymphoma; Transformed Follicular Lymphoma (TFL)
Keywords: CRC01; anti-CD19 CAR-T; CAR-T; CAR T cells; Chimeric antigen receptor; PD-1 knock down; TIGIT knock down
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRC01 (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, CRC01.
  Interventions: Biological: CRC01; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: CRC01 — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells administered intravenously at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg.
Drug: Fludarabine — Administered according to package insert
Drug: Cyclophosphamide — Administered according to package insert

SUMMARY:
This is a multi-center, phase I/II study to determine the efficacy and safety of CRC01 in adult patients with relapsed or refractory large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 19 years of age and provided written informed consent
2. Histologically confirmed following large B-cell lymphomas according to the World Health Organization classification 2017

   * Diffuse large B-cell lymphoma, not otherwise specified Including Large cell transformation from follicular lymphoma (Transformed follicular lymphoma)
   * High-grade B-cell lymphoma, not otherwise specified
   * High-grade B-cell lymphoma with double-hit/triple-hit
   * Primary mediastinal large B cell lymphoma
3. Relapsed or refractory disease after ≥ two lines of chemotherapy including rituximab, anthracycline and either having failed autologous Hematopoietic stem cell transplantation (ASCT) or being ineligible for or not consenting to ASCT.
4. At least one measurable lesion (Long diameter ≥ 1.5cm)
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
6. Adequate renal and hepatic functions based on the laboratory test results

   * Total Bilirubin ≤ 2.0mg/dL with the exception of patients with Gilbert-Meulengracht syndrome; patients with Gilbert-Meulengracht syndrome may be included if their total bilirubin is ≤ 3 X ULN and direct bilirubin ≤ 1.5 X ULN.
   * Aspartate transaminase (AST) and Alanine transaminase (ALT) ≤ 3 X Upper Limit of Normal (ULN) for age with exception of liver metastasis; patients with liver metastasis may be included if their AST and ALT are ≤ 5 X ULN.
   * Serum creatinine ≤ 1.5 X ULN
   * Estimated Glomerular Filtration Rate (eGFR) ≥ 60mL/min/1.73m2
7. Adequate hematologic function without transfusions within 2 weeks prior to screening for the study defined as followings:

   * Hemoglobin > 8.0g/㎗
   * Absolute Neutrophil Count (ANC) > 1,000/㎕
   * Absolute Lymphocyte Count (ALC) ≥ 300/㎕
   * Platelets ≥ 50,000/㎕
8. Must have a minimum level of pulmonary reserve defined as;

   * ≤ Grade 1 dyspnea per Common terminology criteria for adverse events (CTCAE) v5.0
   * pulse oxygenation > 91% on room air
9. Hemodynamically stable, without pericardial effusion and Left Ventricle Ejection Fraction (LVEF) ≥ 50% confirmed by Echocardiogram (ECG) or Multigated Radionuclide Angiography (MUGA)
10. Must have an apheresis product of non-mobilized cells accepted for manufacturing
11. Life expectancy ≥ 12 weeks
12. Women of child-bearing potential and all male participants must agree to use highly effective methods of contraception for at least 12 months following CRC01 infusion and until CRC01 are no longer present by PCR on two consecutive tests

Exclusion Criteria:

1. Patients with the following medical history

   * Previous or concurrent malignancy with the following exceptions:

     * Adequately treated basal cell or squamous cell carcinoma without evidence of recurrence for at least 3 years prior to the study
     * In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to the study
     * A primary malignancy which has been completely resected and in complete remission for ≥ 5 years
   * Unstable angina and/or myocardial infarction within 12 months prior to screening
   * Thromboembolic events, pulmonary embolism or bleeding diatheses within 6 months prior to screening
   * Hypoxemia, significant pleural effusion or significant EKG findings within 6 months prior to the screening
2. Patients with the following concurrent disease at screening:

   * Central Nervous System (CNS) involvement by malignancy by MRI at screening
   * Active infection with hepatitis B (HBsAg positive. But, in case of HBcAb IgG positive, the patient can be enrolled in this study if he/she takes prophylactic anti-viral agent.)
   * Active infection with hepatitis C (HCV RNA positive)
   * Human immunodeficiency virus (HIV) positive
   * Active neurological auto-immune or inflammatory disorder (e.g. Guillain Barre Syndrome, Amyotrophic Lateral Sclerosis)
   * Ventricular tachycardia and atrial fibrillation with rapid ventricular response not controlled with medical treatment within 3 months prior to screening
3. Rapidly progressing the disease as per investigator's discretion
4. Had major surgery requiring general anesthesia or mechanical ventilation within 4 weeks prior to screening (For video-assisted thoracoscopic surgery (VATS) or open-and-closed (ONC) surgery can be applied with within 2 weeks prior to screening.)
5. Severe infection requiring anti-bacterial, anti-fungal or anti-viral medication or uncontrolled active infection
6. The following treatment history is excluded:

   * Prior treatment with any prior anti-CD19/anti-CD3 therapy or any other anti-CD19 therapy
   * Prior treatment with any adoptive T cell therapy
   * Treatment with any prior gene therapy product
   * Prior allogeneic HSCT
   * Patients on oral anticoagulation therapy
7. Eligible for and consenting to ASCT
8. Use of investigational medicinal product/device within 4 weeks prior to screening
9. Pregnant or lactating women
10. Hypersensitivity reaction to the excipients of CRC01 cell product
11. The following treatments are excluded:

    * Anti-neoplastic therapies including chemotherapy, biologic agents, retinoid therapy, radiotherapy, immune therapy, hormonal therapy, etc. other than lymphodepleting chemotherapy within 2 weeks of leukapheresis and within 2 weeks of CRC01 infusion
    * Steroids: therapeutic doses of steroids must be stopped > 7 days prior to leukapheresis and > 5 days prior to CRC01 infusion. However, the following physiological replacement doses of steroids are allowed: < 6 mg/m2/day hydrocortisone or equivalent
    * Immunosuppression: any immunosuppressive medication must be stopped > 4 weeks prior to leukapheresis and > 4 weeks prior to CRC01 infusion
    * Antibody use including anti-CD20 therapy within 4 weeks prior to CRC01 infusion
    * CNS disease prophylaxis must be stopped > 1 week prior to CRC01 infusion (e.g. intrathecal methotrexate)

Other protocol-related inclusion/exclusion may apply.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Study: Maximum Tolerated Dose (MTD) which will be the Recommended Phase 2 Dose (RP2D) | 28 days
Phase 2 Pivotal Study: Overall Response Rate (ORR) | 5 years
  ORR is defined as the incidence of either a complete response (CR) or a partial response (PR) per the Lugano Criteria for Response Assessment (2014).

SECONDARY OUTCOMES:
Time to response (TTR) | 5 years
Duration of overall response (DOR) | 5 years
Event free survival (EFS) | 5 years
Progression free survival (PFS) | 5 years
Overall survival (OS) | 5 years
Incidence and severity of adverse events (AEs) | 5 years
Incidence of immunogenicity to CRC01 | 5 years
Number of participants with presence of exposure to replication-competent lentivirus (RCL) as Assessed by quantitative polymerase chain reaction (qPCR) | 5 years
Incidence of secondary malignancy | 5 years
Peak concentration (Cmax) of CRC01 transduced cells into target tissues | 5 years
Area under the concentration versus time curve (AUC) of CRC01 transduced cells into target tissues | 5 years
Time to maximum observed concentration (Tmax) of CRC01 transduced cells into target tissues | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee YH, Lee HJ, Kim HC, Lee Y, Nam SK, Hupperetz C, Ma JSY, Wang X, Singer O, Kim WS, Kim SJ, Koh Y, Jung I, Kim CH. PD-1 and TIGIT downregulation distinctly affect the effector and early memory phenotypes of CD19-targeting CAR T cells. Mol Ther. 2022 Feb 2;30(2):579-592. doi: 10.1016/j.ymthe.2021.10.004. Epub 2021 Oct 8. PMID 34628052